CLINICAL TRIAL: NCT00807651
Title: Safety and Efficacy Study of Autologous Nonmyeloablative Hematopoietic Stem Cell Transplantation for Early Onset Type 1 Diabetes-a Phase II Study
Brief Title: Autologous Hematopoietic Stem Cell Transplantation for Early Onset Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Guang Ning, Director, Shanghai Jiao Tong University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCEMD006
Record Dates: First submitted 2008-12-11; First posted 2008-12-12 (Estimated); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Diabetes Mellitus; Stem cells; Autologous stem cell transplantation; Autoimmune diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Autoimmune Diseases | interventions — Convulsive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- insulin therapy (Active Comparator): The participants not accepted written informed consent will receive insulin therapy
  Interventions: Drug: Insulin therapy
- AHSCT (Experimental): The participants accepted written informed consent will receive the therapy of autologous hematopoietic stem cell transplantation(AHSCT)
  Interventions: Procedure: AHSCT

INTERVENTIONS:
Procedure: AHSCT — All study participants given written informed consent will perform autologous hematopoietic stem cell transplantation(AHSCT) and be treated with immunosuppression.
  Other Names: hematopoietic stem cell
  Arms: AHSCT
Drug: Insulin therapy — All study participants not accepted written informed consent will received insulin therapy with consistent or multiply subcutaneous injection.
  Other Names: insulin injection therapy
  Arms: insulin therapy

SUMMARY:
This is a phase II trial in individuals who have been diagnosed with type 1 diabetes within the previous 6 months. The study is evaluating whether stem cell transplantation is safe when chemotherapy and immunotherapy are used in combination and if it has immune resetting effect that may halt the immune attack to pancreas islets and thus preserve the body's own insulin production.

DETAILED DESCRIPTION:
Type 1 diabetes is an autoimmune disease in which the immune system mistakenly attacks the insulin-producing beta cells in the pancreas. Generally, at the time someone is diagnosed with type 1 diabetes, not all of a person's beta cells have been destroyed. It's important to preserving the remaining precious beta cells so as to stop the diabetes progression.

The exact mechanism of action of Autologous Hematopoietic Stem Cell Transplantation(AHST) in autoimmune disorders is not fully understood. Preliminary data supported post-AHST immune resetting included an increase in thymus-derived naive T cells, decreased central-memory T cells, increased output of recent thymic emigrants, and recovery of a diverse but distinct T-cell receptor repertoire following AHST. In the patients of type 1 diabetes, decreasing titer of anti-GAD antibody may bring improvement of beta-cell function after intensive immunosuppression. Furthermore, there may exit the possibility of regeneration of beta cells from surviving beta cells or from pancreatic or bone marrow stem cells.

Patients recently diagnosed (less than 6 months) with type 1 diabetes mellitus proved by positive antibody against glutamic acid decarboxylase will be included in this study. Hematopoietic stem cells will be mobilized with cyclophosphamide (2.0 g/m2) and granulocyte colonystimulating factor (10 μg/kg per day) and then collected from peripheral blood by leukapheresis and cryopreserved. The cells were injected intravenously after conditioning with cyclophosphamide (200 mg/kg) and rabbit antithymocyte globulin (4.5 mg/kg). This procedure is performed in isolated rooms at the Bone Marrow Transplantation Unit of Shanghai Ruijin Hospital affiliated to Shanghai Jiao-Tong University School of Medicine. Patients will be discharged from the hospital 1 month after transplantation and continue the follow-ups for 3 years. Patients fitting the inclusion criteria but not agreeing to perform the transplantation are the control group and they will be followed in parallel with transplanted patients.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus diagnosed by clinical/metabolic parameters and positive anti-GAD antibody
* Less than 6 months from diagnosis

Exclusion Criteria:

* Previous diabetic ketoacidosis
* Pregnancy
* Severe psychiatric disorder
* Severe organic impairment (renal, hepatic, cardiac, pulmonary)
* Active infectious disease
* Previous or present neoplastic disease

Ages: 14 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2008-02 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Exogenous insulin dose | 1 month, 3 months, 6 months, 12 months, 24 months, 36 months

SECONDARY OUTCOMES:
Anti-GAD titres | 1 month, 3 months, 6 months, 12 months, 24 months, 36 months
C-peptide level | 1 month, 3 months, 6 months, 12 months, 24 months, 36 months
HbA1c level | 3 months, 6 months, 12 months, 24 months, 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Guang Ning, MD. PhD., Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Voltarelli JC, Couri CE, Stracieri AB, Oliveira MC, Moraes DA, Pieroni F, Coutinho M, Malmegrim KC, Foss-Freitas MC, Simoes BP, Foss MC, Squiers E, Burt RK. Autologous nonmyeloablative hematopoietic stem cell transplantation in newly diagnosed type 1 diabetes mellitus. JAMA. 2007 Apr 11;297(14):1568-76. doi: 10.1001/jama.297.14.1568. PMID 17426276
- [Derived] Ye L, Li L, Wan B, Yang M, Hong J, Gu W, Wang W, Ning G. Immune response after autologous hematopoietic stem cell transplantation in type 1 diabetes mellitus. Stem Cell Res Ther. 2017 Apr 18;8(1):90. doi: 10.1186/s13287-017-0542-1. PMID 28420440
- [Derived] Gu W, Hu J, Wang W, Li L, Tang W, Sun S, Cui W, Ye L, Zhang Y, Hong J, Zhu D, Ning G. Diabetic ketoacidosis at diagnosis influences complete remission after treatment with hematopoietic stem cell transplantation in adolescents with type 1 diabetes. Diabetes Care. 2012 Jul;35(7):1413-9. doi: 10.2337/dc11-2161. PMID 22723579
- [Derived] Zhang X, Ye L, Hu J, Tang W, Liu R, Yang M, Hong J, Wang W, Ning G, Gu W. Acute response of peripheral blood cell to autologous hematopoietic stem cell transplantation in type 1 diabetic patient. PLoS One. 2012;7(2):e31887. doi: 10.1371/journal.pone.0031887. Epub 2012 Feb 22. PMID 22384093